CLINICAL TRIAL: NCT07182136
Title: The Impact of Hepatic Steatosis on Survival After Pancreaticoduodenectomy for Resectable Pancreatic Cancer. A Multifactorial Analysis of Metabolic Dysfunction
Brief Title: The Impact of Hepatic Steatosis on Survival After Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: Wei-Hsun Lu (Other)
Responsible Party: Sponsor-Investigator, Wei-Hsun Lu, MD, National Cheng Kung University
Organization: National Cheng Kung University (Other)
Other Study IDs: ChengKungUniversityTainan
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Nonalcoholic Fatty Liver Disease After Pancreaticoduodenectomy
Keywords: pancreatic ductal adenocarcinoma, pancreaticoduodenectomy, hepatic steatosis, nonalcoholic fatty liver disease, exocrine insufficiency
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pancreaticoduodenectomy — Retrospective study evaluating postoperative NAFLD and metabolic outcomes in patients with stage I-II pancreatic cancer after PD.

SUMMARY:
We will use simple summaries, educational handouts, and discussions with doctors and nurses to explain this study. The study looks at patients with early-stage pancreatic cancer who undergo pancreaticoduodenectomy (Whipple surgery). We found that some patients develop fatty liver (non-alcoholic fatty liver disease, NAFLD) within six months after surgery, which can affect nutrition, blood sugar control, and long-term survival.

To help patients and families understand, we will:

1. Provide clear written information sheets about the purpose of the study and its findings.
2. Use diagrams or plain-language explanations of terms like "pancreatic exocrine function" and "fatty liver."
3. Share results with healthcare providers so they can guide patients in nutrition, enzyme replacement, diabetes monitoring, and follow-up care.
4. Offer contact information for the research team to answer questions.

ELIGIBILITY:
Inclusion Criteria:

* Adults with stage I-II pancreatic ductal adenocarcinoma.
* Underwent curative-intent pancreaticoduodenectomy (conventional or pylorus-preserving).
* Surgery between January 2015 and May 2023.
* Complete clinical and imaging data available.
* Survived at least 6 months postoperatively.

Exclusion Criteria:

* Preoperative hepatic steatosis
* Incomplete clinical or imaging data
* Death within 6 months after surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Two hundred patients with stage I-II pancreatic ductal adenocarcinoma who underwent pancreaticoduodenectomy between 2015 and 2023 at two Taiwanese tertiary centers were included; those with preoperative fatty liver, incomplete data, or early death were excluded
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nonalcoholic fatty liver disease (NAFLD) | 6 months after pancreaticoduodenectomy